CLINICAL TRIAL: NCT05986474
Title: Development of Synthetic Medical Data Generation Technology to Predict Postoperative Complications
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hajeong Lee, Associate Professor, Seoul National University Hospital
Other Study IDs: H-2102-192-1203
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acute Kidney Injury; Surgery-Complications; Nephropathy
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
<Development of synthetic medical data generation technology to predict postoperative complications>

In order to develop a model for predicting the occurrence of complications after surgery, it is necessary to establish a cohort along with statistical indicators related to the occurrence of complications. This study aims to combine synthetic medical data based on actual clinical data and develop a predictive model based on synthetic medical data.

This will allow researchers to conduct research only with synthetic data without dealing with actual medical data, allowing them to use and process data without legal constraints, and to create as much data as they want based on various preprocessed, standardized, and labeled raw data.

Patients from three hospitals in Korea (Seoul National University Hospital, Seoul National University Bundang Hospital, Seoul Metropolitan City-Boramae Medical Center) were enrolled for the study.

Medical data (both clinical and laboratory) from 410,000 patients who were conducted surgery between 2005 and 2020 were collected to evaluate the performance of the prediction model using AKI-based prediction model development and external verification.

Based on the collected patient data, synthetic medical data were combined using the machine learning algorithm, and the anonymity and re-identification of the synthesized medical data were evaluated.

Also, the development of AI-based prediction model using synthetic medical data and the actual medical data model were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years.
* Non-cardiothoracic and non-vascular surgery from five departments (general surgery, obstetrics and gynecology (OBGY), urologic surgery, neurosurgery, and orthopedic surgery)

Exclusion Criteria:

* 1) no information of baseline (≤90 days before surgery) or follow-up (≤7 days after surgery) renal function
* 2) exclusive surgery, including surgeries of deceased patients or surgery that directly affect renal function (partial or total nephrectomy, kidney transplantation)
* 3) preoperative advanced kidney dysfunction, including preoperative serum creatinine (SCr) ≥4.0 mg/dL, baseline eGFR (estimated glomerular filtration rate) <15 mL/min/1.73 m2, preoperative kidney replacement therapy history, or AKI history within 2 weeks of surgery
* 4) surgery other than general or spinal anesthesia (local anesthesia or monitored anesthesia care)
* 5) missing covariates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years who underwent non-cardiothoracic and non-vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 410000 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | After surgery, within 7 days
  Surgical complication 1
Acute kidney disease | After surgery, within 3 months
  Surgical complication 2

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho JM, Kwon S, Yang S, Park J, Jeong S, Park S, Ryu J, Kim S, Lee J, Lee JP, Yoon HJ, Kim DK, Joo KW, Kim YS, Kim K, Park M, Lee H. Acute kidney injury after non-cardiac major surgery: has it reduced? Clin Kidney J. 2024 Jun 19;17(7):sfae183. doi: 10.1093/ckj/sfae183. eCollection 2024 Jul. PMID 39831175